CLINICAL TRIAL: NCT00351026
Title: Methadone Maintenance & HIV Risk in Ukraine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R21DA021073 (NIH); R21DA021073 (NIH)
Record Dates: First submitted 2006-07-10; First posted 2006-07-12 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Opioid Dependence
Keywords: opioid dependence; methadone; HIV
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Methadone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): 25 HIV negative opiate dependent patients all treated with methadone
  Interventions: Drug: Methadone
- 2 (Active Comparator): 25 HIV positive opiate dependent patients all treated with methadone
  Interventions: Drug: Methadone

INTERVENTIONS:
Drug: Methadone — short-term methadone maintenance

SUMMARY:
Treatment of opioid dependence is an important way to reduce the spread of HIV and other infectious diseases, particularly in Ukraine since intravenous opioid use is the major way these infections are being spread. This proposal will be done at the Kiev City Narcology Hospital and the City AIDS Center with collaborators from the University of Alabama and the University of Colorado. It will study the acceptability and impact of a 3-month course of methadone maintenance on 50 persons with opioid dependence, 25 who are HIV+ and 25 HIV-. The proposed work will build on a relationship that was established with the Ukrainian Co-Principal Investigator, Sergiy Dvoryak, M.D., during his Humphrey Fellowship at Johns Hopkins in 1999-2000 when he spent time with Dr. Woody and Metzger at the Penn Addiction and Treatment and Research Center. It will also extend studies of pharmacologic treatment for opioid dependence and risk reduction behavioral interventions that are being done by Drs. Woody, Schumacher and Booth in Russia and Ukraine. Primary aims are to: measure the acceptability and compliance with a 3-month course of methadone maintenance in HIV+ and HIV- patients; measure the impact of a 3-month course of methadone in reducing opioid use in HIV+ and HIV- patients; measure the impact of a 3-month course of methadone on reducing HIV risk behavior in HIV+_and HIV- patients. Secondary aims are to: assess the degree to which a 3-month course of methadone maintenance reduces illegal activities and improves employment and psychiatric symptoms; determine short-term outcome after completion of methadone treatment; and obtain pilot data on the prevalence of hepatitis B and C among study patients. This study will provide pilot data on the acceptability and efficacy of a short-term course of methadone maintenance on HIV+ and HIV- persons in a setting where this treatment has not been evaluated, on the feasibility of conducting the kind of work that is proposed, and will enhance research capabilities of Kiev investigators for future HIV prevention and treatment studies.

DETAILED DESCRIPTION:
Approximately 40 subjects have been enrolled in this study as of September 1, 2009. Almost all have completed the 12 week study period and elected to transfer to the regular methadone program at the same location, that was started in the last 2 years with support from the Global Fund. A 1-year supplement has been awarded to pilot test an intervention developed by Dr. Dvoryak to facilitate enrollment in methadone by persons who could benefit, and an intervention called "Life Steps" developed by Safren and colleagues and aimed to facilitate adherence to antiretroviral therapy. A site visit was completed in 5/09 in which we conducted two focus groups to determine local conditions that needed to be included in Life Steps so as to make it relevant to Ukrainian cultural conditions, followed by modification and training in the slightly revised version of Life Steps. We anticipate that the 25 additional HIV+ patients who will be enrolled to complete the supplement will start to be enrolled in 10/09, when recruitment for the parent study has been completed.

ELIGIBILITY:
Inclusion Criteria:

Primary diagnosis of current opioid dependence with physiological features, present for at least one year and seeking outpatient treatment.

Age between 18 and 40 Stable address within Kiev and not planning to move Home telephone number where can be reached Willingness and ability to give informed consent and otherwise participate

Exclusion Criteria:

Clinically significant cognitive impairment, schizophrenia, paranoid disorder, bipolar disorder, or seizure disorder Advanced neurological, cardiovascular, renal, hepatic or other medical disorder that would seriously impair or make hazardous patient's ability to participate Active tuberculosis Currently dependent on alcohol, benzodiazepines or other sedative-like drugs Pending legal charges with potential impending incarceration Plans to move from the area within the next 6 months Concurrent participation in another treatment study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-06; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Measure the acceptability and compliance with a 3-month course of methadone maintenance in HIV+ and HIV- patients in this cultural setting | 3 months
Measure the impact of a 3-month course of methadone treatment in HIV+ and HIV- on reducing opioid use | 3 months
Measure the impact of a 3-month course of methadone treatment in HIV+ and HIV- on reducing HIV risk behavior | 3 months

SECONDARY OUTCOMES:
Assess the degree to which the 3-month course of methadone maintenance reduces illegal activities and improves employment and psychiatric symptoms | 3 months
Determine short term outcome after completion of methadone treatment | 3 months
Obtain pilot data on the prevalence of hepatitis B and C among study patients | 3 months

CONTACTS AND LOCATIONS:
Locations (2):
- Ukraine (2):
  - Kiev City AIDS Center, Kiev
  - City AIDS Center, Kiev